CLINICAL TRIAL: NCT06085131
Title: Accuracy of the New Barrett TAL Formula With the Argos Measurements: A Multicenter Prospective Study
Status: Completed | Type: Observational
Sponsor: Shammas Eye Medical Center (Other)
Collaborators: Sengi (Industry)
Responsible Party: Sponsor
Other Study IDs: HJS-23-01
Record Dates: First submitted 2023-10-10; First posted 2023-10-16 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Argos Biometer: Preoperative biometry with the Argos device
  Interventions: Device: Argos

INTERVENTIONS:
Device: Argos — Argos Biometer

SUMMARY:
This study is a prospective, multi-site, multi-surgeon, observational study of refractive accuracy with the Argos using BTAL after successful cataract surgery. Subjects will be assessed pre-operatively, operatively and at 5-8 weeks postoperatively. Clinical evaluations will include measurement of visual acuity, manifest refraction, and preoperative biometry.

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible for the study if they meet the following criteria:

* Cataract surgery that was completed without complications with biometry measured using the Argos biometer.
* Subjects that elect Clareon SY60WF aspheric lens (Alcon, Fort Worth, TX).
* Potential post-operative visual acuity of better than logMAR 0.30 (20/40).
* BTAL was used to determine the IOL power implanted.

Exclusion Criteria:

If any of the following exclusion criteria are applicable to the subject or either eye, the subject should not be enrolled in the study.

* Patients with pre-existing ocular pathology that in the opinion of the principial investigator would influence the postoperative refraction.
* Any disease or pathology, including but not limited to irregular corneal astigmatism and keratoconus, that is expected to reduce the potential postoperative BCDVA to a level worse than 20/40.
* Patients with history of previous ocular surgery.
* Patients with signs of inability to understand consent for study and procedure planned.
* Eyes with intraoperative or postoperative complications.
* Suboptimal surgical outcomes that are not related to the treatment plan, e.g. capsular tear, cystoid macular edema.
* Astigmatism >±0.75D.

Each investigator reserves the right to declare a patient ineligible or non-evaluable based on medical evidence that indicates they are unsuitable for the trial.

Pregnancy has a known effect on the stability of refractions and visual acuity. As such, subjects who become pregnant during the study will not be discontinued but their data may be excluded from analyses of effectiveness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible test subjects will be adults who are interested in and appropriate candidates for cataract surgery.
Sampling Method: Non-Probability Sample
Enrollment: 501 (Actual)
Dates: Start 2023-10-31 (Actual); Primary Completion 2025-01-29 (Actual); Study Completion 2025-01-29 (Actual)

PRIMARY OUTCOMES:
The percentage of eyes that achieve a postoperative manifest spherical equivalent refraction ≤ ±0.50 D. | 2 months postoperative

SECONDARY OUTCOMES:
The percentage of eyes that achieve a postoperative manifest spherical equivalent refraction ≤ ±0.250D, ≤ ±0.75D and ≤ ±1.00D. | 2 months postoperative
The Mean Predictive Error and its standard deviation after constant personalization for the entire series. | 2 months postoperative
The Mean Predictive Errors in the short eyes and in the long eyes | 2 months postoperative
  The Mean Predictive Errors in the short eyes and in the long eyes (Short AL<22.5mm, Long AL >24.5mm and Medium AL 22.6mm to 24.4mm), and the percentage of eyes that achieve a postoperative manifest spherical equivalent refraction ≤ ±0.25 D, ≤ ±0.50 D, ≤ ±0.75 D and ≤ ±1.00 D in each of these categories.

CONTACTS AND LOCATIONS:
Overall Officials: H J Shammas, MD, Principal Investigator — Shammes Eye Medical Center
Locations (6):
- United States (6):
  - Colvard-Kandavel Eye Center, Encino, California
  - Shammas Eye Medical Center, Lynwood, California
  - Shammas Eye Center, Whittier, California
  - Multack Eye Care, Sc, Frankfort, Illinois
  - Multack Eye Care, SC, Olympia Fields, Illinois
  - Juliette Eye Institute, Albuquerque, New Mexico